CLINICAL TRIAL: NCT04769245
Title: The Effectiveness of ACB-IP 1.0 Universal Pathogen Free Concentrated Cocktail Convalescent Plasma in COVID-19 Infection
Brief Title: The Effectiveness of ACB-IP 1.0 Convalescent Plasma in COVID-19 Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Acibadem University (Other)
Collaborators: Acıbadem Labcell (Other)
Responsible Party: Sponsor
Other Study IDs: Acibadem Healthcare Group
Record Dates: First submitted 2021-02-15; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Single donor convalescent plasma: Patients who had positive reverse-transcriptase-polymerase-chain-reaction (RT-PCR) for SARS-CoV2 and radiologically confirmed pneumonia treated with single donor plasma
- ACB- IP 1.0: Patients who had positive reverse-transcriptase-polymerase-chain-reaction (RT-PCR) for SARS-CoV2 and radiologically confirmed pneumonia treated with ACB- IP 1.0 pathogen-free concentrated cocktail convalescent plasma

SUMMARY:
Pathogen-free, concentrated, pooled convalescent plasma has higher SARS-CoV2 antibody titers and neutralizing antibody activities, without requiring blood group compatibility that allows patient accessibility in a shorter time and has safe plasma characteristic.

DETAILED DESCRIPTION:
The efficacy of SARS-CoV2 standard single donor convalescent plasma varied according to the application time and most importantly the amount of antibody that is administered. Single donor plasma has some drawbacks; such as the insufficient levels of neutralizing antibody activities, the requirements of blood group compatibility, and the risk of infection transmission. In this study, the efficacy and safety of pathogen inactivated, isohemagglutinin-depleted (concentrated) and pooled convalescent plasma was investigated.

ELIGIBILITY:
Inclusion Criteria:

* Are over the age of 60 or-
* Between the ages of 18-60, serious comorbidities (cancer, COPD, cardiovascular illness, hypertension, DM)
* Clinically diagnose COVID-19 or radiological diagnosed COVID-19 pnemonia

Exclusion Criteria:

* Multiple Organ Failure

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults with positive reverse-transcriptase-polymerase-chain-reaction (RT-PCR) for SARS-CoV2 and/or radiologically confirmed pneumonia, were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-02-18 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Mortality Rate | 6 Months
  A mortality rate is a measure of the frequency of occurrence of death in a defined population during a specified interval.
Length of Hospitalization | 6 Months
  The average length of stay in hospitals (ALOS) is often used as an indicator of efficiency

SECONDARY OUTCOMES:
Side Effects | 6 Months
  Problems that occur when treatment goes beyond the desired effect. Or problems that occur in addition to the desired therapeutic effect.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Acıbadem Labcell Cellular Therapy Laboratories, Istanbul
  - Acibadem Altunizade Hospital, Istanbul